CLINICAL TRIAL: NCT03365271
Title: Study on the Post-operative Effect of Applying Drainage on Total Knee Arthroplasty
Brief Title: The Post-operative Effect of Applying Drainage on Total Knee Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Lin Chutong, The clinical professor of arthritis clinic and research center, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PUPHEMS
Record Dates: First submitted 2017-11-25; First posted 2017-12-07 (Actual); Last update posted 2017-12-07 (Actual); Status verified 2017-12

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Drainage

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- drainage (Experimental): A drainage will be applied in this group.
  Interventions: Procedure: drainage
- without drainage (Active Comparator): Non-drainage will be applied in this group.
  Interventions: Procedure: non-drainage

INTERVENTIONS:
Procedure: drainage — Applying a drain tube during TKA procedure
  Arms: drainage
Procedure: non-drainage — No drain tube will be applied during TKA procedure
  Arms: without drainage

SUMMARY:
This multicenter clinical trial aims to investigate the exact effect of drainage use for osteoarthritis patients in total knee arthroplasty (TKA) on post-operative performance.

DETAILED DESCRIPTION:
This is a multicenter,open-label randomized controlled trail. A total of 100 participants will receive same perioperative treatment schedule, and all surgeries will be carried out by the same surgeon. Among all the participants, 50 patients will be randomly assigned to the experiment group in which a drainage will be applied during the surgery, while another 50 patients will be randomly assigned to the control group without a drainage application in the surgery.Data on perioperative bleeding volume, swelling of lower extremities, pain score will be collected and analysed.

ELIGIBILITY:
Inclusion Criteria:

* Ready to receive single-side TKA
* Be evaluated as ASA 1-2 degree before operation

Exclusion Criteria:

* coagulation disorder
* peripheral vessel diseases
* contraindication of surgery

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-02 (Estimated); Primary Completion 2018-08 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
The change of bleeding volume in perioperative period | before operation and one week after operation
  The difference between baseline Hct collected before operation and Hct collected one week after operation

SECONDARY OUTCOMES:
Swelling of the lower extremities | one week after operation
  perimeter of lower extremities before and after operation
Range of motion | one week after operation
  Range of motion of the knee received operation
Pain | one week after operation
  Use the Visual Analogue Scale to estimate the pain and its score ranges from 0 to 10. The higher the score is, the more severe pain the patient is feeling.

CONTACTS AND LOCATIONS:
Overall Officials: Jianhao Lin, MD, Principal Investigator — arthritis clinic and research center